CLINICAL TRIAL: NCT05306132
Title: A Phase I ,Open, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of ASKC202 With or Without ASK120067 in Patients With Advanced Solid Tumors
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of ASKC202 With or Without ASK120067
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASKC202-001
Record Dates: First submitted 2022-03-23; First posted 2022-03-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASKC202 (Experimental): Participants received ASKC2020 50mg~600mg orally
  Interventions: Drug: ASKC202
- ASKC202 plus ASK120067 (Experimental): Participants received ASKC202 150 mg or 200 mg qd orally plus ASK120067 80 mg bid orally
  Interventions: Drug: ASKC202; Drug: ASK120067

INTERVENTIONS:
Drug: ASKC202 — Dosage Forms: Tablets; Administration: Oral administration
Drug: ASK120067 — Dosage Forms: Tablets; Administration: Oral administration
  Other Names: Limertinib
  Arms: ASKC202 plus ASK120067

SUMMARY:
This study is the first-in-human of ASKC202, which is an open-label, non-randomized, multicenter study with a dose escalation phase and a dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed and dated informed consent;
2. Aged 18 years old or more, male or female;
3. Part 1 (Monotherapy Dose-Escalation) and Part 3 (Monotherapy Expansion): the subjects with locally advanced or metastatic solid tumors for whom no standard therapy regimens are available currently or who are intolerable to standard therapy regimens; Part 3: the subjects with MET gene amplification or protein overexpression; Part 3 cohort 1: histologically or cytologically confirmed unresectable locally advanced or metastatic NSCLC.

4）Part 2:(Combination Therapy Dose-Escalation):a)histologically or cytologically confirmed unresectable locally advanced or metastatic NSCLC;b)Histologically confirmed EGFR sensitizing mutation (Ex19del or L858R).；c)Disease progression following treatment with a third-generation EGFR TKI, or treatment with a first-/second-generation EGFR-TKI with confirmed T790M-negative status upon progression; d)MET gene amplification or protein overexpression.

5) Part 4:(Combination Therapy Dose-Expansion):a)histologically or cytologically confirmed unresectable locally advanced or metastatic NSCLC;b)Histologically confirmed EGFR sensitizing mutation (Ex19del or L858R).；c)MET gene amplification or protein overexpression.

6) At least one measurable lesion (based on the RECIST 1.1 criterion) (this article is only for the dose expansion phase); 7) ECOG score 0~1; 8) Expected survival time ≥ 3 months; 9) Major organ function is essentially normal (no transfusions, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), or other medically supportive care have been received in the 14 days prior to the administration of the study drug), and laboratory tests during the screening period meet the following criteria: system Laboratory test values haematology Absolute neutrophil count ≥1.5 ×109/L platelet ≥90×109/L haemoglobin ≥90g/L kidney Serum creatinine or Creatinine clearance (CrCl). ≤ 1.5 × ULN or

≥60 mL/min (estimated from the Cockcroft-Gault formula) liver Total bilirubin ≤1.5 × ULN or ≤2 × ULN (for patients with liver cancer or liver metastases). AST(SGOT) and ALT (SGPT). ≤2.5 × ULN or ≤5 × ULN (for patients with liver cancer or liver metastases). Coagulation (no anticoagulation was received in the 7 days prior to the administration of the study drug).

International normalized ratio (INR) or prothrombin time (PT). ≤1.5 × ULN Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN 10) Women of childbearing age must have a pregnancy test (serum or urine) within 7 days of enrolling and have a negative result, or meet one of the following criteria to prove that there is no risk of pregnancy: a Postmenopausal is defined as amenorrhea at least 12 months after age >50 years and discontinuation of all exogenous hormone replacement therapy; b Women younger than 50 years of age who are considered postmenopausal if they have been amenorrhea for 12 months or more after stopping all exogenous hormone therapy, and luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within the laboratory reference values for postmenopausal; c Previously undergone irreversible sterilization procedures, including hysterectomy, bilateral ovarian resection, or bilateral salping, with the exception of bilateral tubal ligation; 11) Women of childbearing age should use strict contraceptive contraception throughout trial 7 and within 3 months after the last dose of the test drug; male subjects should use strict contraception throughout the trial period and for 6 months after the last dose of the test drug and no sperm donation; 12) The patient understands the purpose and steps of the trial, voluntarily participates in the trial, and signs a written informed consent form; 13) Patients have good comprehension, are able to follow protocol requirements and can cooperate with investigators in this trial.

Exclusion Criteria:

1. Have previously received or are receiving any treatment for c-Mets (including all monoclonal antibodies or small molecule drugs targeted at the target, except for crizotinib);
2. Have received chemotherapy, hormone therapy, immunotherapy, or biological therapy such as antibody therapy within 4 weeks prior to the first dose, or traditional Chinese medicine with anti-tumor indications within 2 weeks, or small molecule targeted therapy with an interval of less than 5 half-lives; palliative radiotherapy within 7 days or extensive/therapeutic radiotherapy within 14 days prior to the first dose;
3. Those who still need to continue to use systemic immunosuppressants or systemic corticosteroids (≥ 10 mg of prednisone or its equivalent other corticosteroid) for 2 weeks prior to the first dose;
4. Patients who have used strong inhibitors or strong inducers of CYP3A within 2 weeks prior to the first administration, or who need to continue treatment with these drugs during the study period;
5. Participation in clinical trials of other drugs within 4 weeks prior to the first administration (except for failed screening);
6. Patients who underwent other major surgical procedures other than diagnosis or biopsy within 4 weeks prior to the first dose, or who were expected to undergo major surgeries during the study period;
7. Prior to the first administration, there are unhealed toxic reactions of ≥ grade 2 (CTCAE 5.0 standard) associated with any previous treatment, any level of hair loss, and platinum drugs Except for grade 2 neuropathy caused;
8. Patients with primary central nervous system tumors or central nervous system metastases including meningeal metastases (except those who are asymptomatic and stable, do not require steroid use for at least 4 weeks before the first dose);
9. Gastrointestinal disorders (e.g., Crohn's disease, ulcerative colitis, intestinal obstruction, short bowel syndrome) or other malabsorption conditions that have difficulty swallowing or affect drug absorption;
10. There are any other serious or uncontrolled acute and chronic diseases, such as severe or uncontrollable liver or kidney disease (except liver and kidney cancer), uncontrollable hypertension (blood pressure > 150/95 mmHg after antihypertensive therapy), and Acute pancreatitis, uncontrollable hyperglycemia (fasting blood glucose >8.0 mmol/L after hypoglycemic therapy), severe or uncontrolled eye lesions, etc
11. Previous history includes interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid therapy, or evidence of clinically active ILD
12. Have previously received hematopoietic stem cell transplants or solid organ transplants, or plan to receive hematopoietic stem cell transplants or solid organ transplants during the current period of study;
13. If not controlled, large pleural effusions, pericardial effusions, or ascites that need to be drained still need;
14. There are serious or active infections that required intravenous antibiotics or hospitalization, such as HBV (HBsAg-positive and peripheral HBV-DNA titer test≥1×10^4 copies/mL or 2000 IU/mL), HCV, HIV, and syphilis
15. Meets any of the following cardiac criteria:

    a Average QTc interval prolongation of 3 ECG examinations at rest (QTcF: 450 ms> for men > 470 ms for women, corrected by Fredericcia's formula); b Presence of uncontrolled or symptomatic arrhythmias, familial arrhythmias, or congenital long QT syndromes; c Had undergone coronary angioplasty, stent implantation, and coronary artery bypass grafting within 6 months before admission; d Myocardial ischemia or myocardial infarction, unstable angina within 6 months before admission; e Judged to be class III-IV congestive heart failure according to the New York Heart Association's cardiac function grade; f Echocardiography (ECHO) shows a left ventricular ejection fraction (LVEF) ≤ 50%;
16. allergies, or a previous history of severe allergies, or known allergies to any of the components of the drug under study;
17. Pregnant, Lactating women;
18. Other primary malignancies have been diagnosed within the last 5 years, and the following conditions can be enrolled: non-melanoma skin cancer, superficial bladder cancer, cervical carcinoma in situ that has undergone surgery and has been cured;
19. Alcohol abuse, substance abuse, and other conditions that may increase the risk of the study or may interfere with study execution and analysis of results, or that the investigator believes that there are other reasons for which they are not suitable for this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and case number of DLT (Dose Limiting Toxicity) during observation period | up to 21 days following first dose
  DLT is short for Dose Limiting Toxicity，dose-limiting describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Maximum Tolerated Dose (MTD） | up to 21 days following first dose
  The MTD was defined as the highest dose of ASKC202 not causing DLT in more than 33% of patients in the first treatment cycle.
Number of participants with adverse events and serious adverse events as assessed by CTCAE v5.0 | up to 30 days following last dose
  An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs. Number of Participants with TEAEs and serious TEAEs were reported.

SECONDARY OUTCOMES:
Pharmacokinetics:maximum Plasma Concentration [Cmax] | up to 21 days following first dose
  Serum samples will be collected for Cmax analysis.
Pharmacokinetics:terminal elimination half life (T1/2) | up to 21 days following first dose
  Serum samples will be collected for T1/2 analysis.
Pharmacokinetics:Area Under Curve (AUC) | up to 21 days following first dose
  Serum samples will be collected for AUC analysis.
ORR | through study completion, an average of 2 years
  Objective response rate (ORR) is defined as the percentage of complete response (CR) or partial response (PR), as determined according to RECIST v1.1.
DCR | through study completion, an average of 2 years
  Disease control rate (DCR) is defined as the percentage of CR or PR or stable disease (SD) , as determined according to RECIST v1.1.
DepOR | through study completion, an average of 2 years
  Depth of response (DepOR) is defined as the maximum percentage change in tumor size compared with baseline.
PFS | through study completion, an average of 2 years
  Progression-free survival (PFS) is defined as the time from the date of first treatment to the first occurrence of disease progression or death from any cause (whichever comes first), as determined according to RECIST v1.1.
DOR | through study completion, an average of 2 years
  Duration of response (DOR) is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever comes first), as determined according to RECIST v1.1.
OS | through study completion, an average of 3 years
  overall survival (OS) is defined as the time from the date of first treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Caicun, MD, Principal Investigator — Shanghai East Hospital Affiliated to Tongji University
Locations (3):
- China (3):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Shanghai East Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No